CLINICAL TRIAL: NCT04247204
Title: 3D Power Doppler Ultrasound Assessment of Endometrial and Sub-endometrial Vascularity Before and After PRP Infusion in Frozen-thawed Embryo Transfer Cycles: a Pilot Study.
Brief Title: Assessment of Endometrial and Sub-endometrial Vascularity Before and After PRP Infusion in Frozen Embryo Transfer Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hatem AbuHashim (Other)
Responsible Party: Sponsor-Investigator, Hatem AbuHashim, Professor, Mansoura University
Organization: Mansoura University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R.20.01.711
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Frozen Embryo Transfer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Platelet-rich plasma (PRP) intrauterine infusion (Experimental)
  Interventions: Biological: Platelet-rich plasma intrauterine infusion

INTERVENTIONS:
Biological: Platelet-rich plasma intrauterine infusion — For all women, basic transvaginal sonography will be done in the 2nd day of frozen embryo transfer (FET) cycle and they will receive standard hormone replacement therapy (HRT) in the form of estradiol valerate tablets (white tablets of Cyclo-Progynova; Bayer Schering Pharma AG, Germany) at a dose of 4mg for 7 days then 6mg for 6 days. Endometrial assessment will be done on day 15 of FET cycle. Those with endometrial thickness between 8-14 mm will be evaluated for endometrial and sub-endometrial vasculature pattern by 3D power Doppler analysis. Then 1 ml of PRP (prepared from autologous blood) will be infused in the uterine cavity and vaginal progesterone 400 mg twice daily will be prescribed for 3 days. Subsequently, D3 embryos will be transferred. Endometrial, sub-endometrial and uterine arterial vascularity pattern will be re-evaluated on the day of ET. Both estradiol valerate tablets and vaginal progesterone will be continued up to 12th week of gestation in case of pregnancy.

SUMMARY:
A good quality embryo and receptive endometrium are important aspects in achieving optimal outcomes in assisted reproductive treatment (ART). Endometrial thickness is an important marker of uterine receptivity. A thin endometrium defined by an endometrial thickness ≤7mm was reported as a poor factor associated with significantly lower implantation and pregnancy rates as well as a higher risk of miscarriage.

Nowadays, platelet-rich plasma (PRP) intrauterine infusion is a promising approach for the treatment of refractory thin endometrium in patients undergoing frozen-thawed embryo transfer. This is based on its ability to stimulate proliferation and angiogenesis with a large number of growth factors and cytokines i.e. the endometrium becomes thicker, with higher vascularity. PRP is easily prepared from an autologous blood sample that eliminates the risk of immunological reactions and transmission infections at low cost.

Endometrial blood flow is another important marker reflective of uterine receptivity. Although publications are increasing concerning the efficacy of PRP intrauterine infusion on endometrial expansion and proliferation in frozen-thawed embryo transfer cycles, yet its angiogenetic effects have not been evaluated so far in either thin endometrium or normal endometrium thickness.

Our study aims to evaluate endometrial and sub-endometrial vasculature patterns before and after PRP infusion in frozen-thawed embryo transfer cycles with normal endometrium thickness.

ELIGIBILITY:
Inclusion Criteria:

* Subfertile women undergoing frozen-thawed embryo transfer with at least previously failed one ICSI cycle.
* Age between 20-35 years.
* Women with endometrium thickness between 8-14 mm on D15 of the frozen embryo transfer cycle

Exclusion Criteria:

* Women with a thin endometrium (≤ 7 mm) on day 15 of the cycle.
* Women with known hematological or immunological disorders
* Women with uncontrolled endocrine or other medical conditions, such as hyperprolactinemia or thyroid diseases.
* Women with uterine abnormalities e.g. Asherman syndrome, myomas, uterine septum, bicornuate uterus.
* Women who refuse to participate in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-08 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-10-05 (Estimated)

PRIMARY OUTCOMES:
Vascularization index of the endometrial region | Day 15 to 18 of the frozen embryo transfer cycle
  Vascularization index of the endometrial region will be measured by a researcher using the built-in VOCAL (Virtual Organ Computer-Aided Analysis) software for 3D power Doppler analysis.

SECONDARY OUTCOMES:
Flow index of the endometrial region | Day 15 to 18 of the frozen embryo transfer cycle
  Flow index of the endometrial region will be measured by a researcher using the built-in VOCAL (Virtual Organ Computer-Aided Analysis) software for 3D power Doppler analysis
Vascularization flow index of the endometrial region | Day 15 to 18 of the frozen embryo transfer cycle
  Vascularization flow index of the endometrial region will be measured by a researcher using the built-in VOCAL (Virtual Organ Computer-Aided Analysis) software for 3D power Doppler analysis
Vascularization index of the sub-endometrial region | Day 15 to 18 of the frozen embryo transfer cycle
  Vascularization flow index of the sub-endometrial region will be measured by a researcher using the built-in VOCAL (Virtual Organ Computer-Aided Analysis) software for 3D power Doppler analysis
Flow index of the sub-endometrial region | Day 15 to 18 of the frozen embryo transfer cycle
  Flow index of the sub-endometrial region will be measured by a researcher using the built-in VOCAL (Virtual Organ Computer-Aided Analysis) software for 3D power Doppler analysis
Vascularization flow index of the sub-endometrial region | Day 15 to 18 of the frozen embryo transfer cycle
  Vascularization flow index of the sub-endometrial region will be measured by a researcher using the built-in VOCAL (Virtual Organ Computer-Aided Analysis) software for 3D power Doppler analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hatem Abu Hashim, MD. FRCOG. PhD, Study Chair — Faculty of Medicine, Mansoura University; Mohamed Taman, MD, Principal Investigator — Faculty of Medicine, Mansoura University

REFERENCES:
- [Background] Nandi A, Martins WP, Jayaprakasan K, Clewes JS, Campbell BK, Raine-Fenning NJ. Assessment of endometrial and subendometrial blood flow in women undergoing frozen embryo transfer cycles. Reprod Biomed Online. 2014 Mar;28(3):343-51. doi: 10.1016/j.rbmo.2013.11.004. Epub 2013 Nov 22. PMID 24447958